CLINICAL TRIAL: NCT04750083
Title: A Phase II/III Study Comparing HX008 (a Humanized Monoclonal Antibody Against PD-1) Plus Chemotherapy With Pembrolizumab Plus Chemotherapy as the First-line Treatment in Participants With Advanced or Metastatic Nonsquamous Non-small Cell Lung Cancer.
Brief Title: HX008 Plus Chemotherapy VS Pembrolizumab Plus Chemotherapy As the First-line Treatment in Participants With Advanced or Metastatic Nonsquamous Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taizhou Hanzhong biomedical co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: HX008-NSCLC-II/III-01
Record Dates: First submitted 2021-02-03; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Nonsquamous Non-small Cell Lung Cancer
MeSH Terms: interventions — pembrolizumab; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Who Masked: Participant
Masking Description: Phase II is open-labelled with one arm, and phase III is single-blinded for the participants with 2 arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- phase II (Experimental): Thirty-sixty participants will receive HX008 200 mg intravenously (IV) PLUS pemetrexed 500 mg/m^2 IV PLUS cisplatin 75 mg/m^2 IV OR carboplatin Area Under the Curve (AUC) 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by pembrolizumab 200 mg IV PLUS pemetrexed 500 mg/m^2 IV Q3W for another 31 cycles.
  Interventions: Drug: HX008; Drug: pemetrexed; Drug: cisplatin/carboplatin
- phase III-experimental (Experimental): Three hundred and twenty participants will receive HX008 200 mg intravenously (IV) PLUS pemetrexed 500 mg/m^2 IV PLUS cisplatin 75 mg/m^2 IV OR carboplatin Area Under the Curve (AUC) 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by pembrolizumab 200 mg IV PLUS pemetrexed 500 mg/m^2 IV Q3W for another 31 cycles.
  Interventions: Drug: HX008; Drug: pemetrexed; Drug: cisplatin/carboplatin
- phase III-control (Experimental): Three hundred and twenty participants will receive pembrolizumab 200 mg intravenously (IV) PLUS pemetrexed 500 mg/m^2 IV PLUS cisplatin 75 mg/m^2 IV OR carboplatin Area Under the Curve (AUC) 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by pembrolizumab 200 mg IV PLUS pemetrexed 500 mg/m^2 IV Q3W for another 31 cycles.
  Interventions: Drug: Pembrolizumab; Drug: pemetrexed; Drug: cisplatin/carboplatin

INTERVENTIONS:
Drug: HX008 — HX008 200 mg intravenously (IV) on Day 1 of every 3-week cycle (Q3W) for up to 35 cycles
  Arms: phase II; phase III-experimental
Drug: Pembrolizumab — Pembrolizumab 200 mg intravenously (IV) on Day 1 of Q3W for up to 35 cycles
  Arms: phase III-control
Drug: pemetrexed — pemetrexed 500 mg/m^2 IV on Day 1 of Q3W for up to 35 cycles
Drug: cisplatin/carboplatin — cisplatin 75 mg/m^2 IV OR carboplatin AUC 5 IV on Day 1 of Q3W for 4 cycles

SUMMARY:
This a phase II-III study. In the single-armed phase II period, HX008, a monoclonal antibody targeting PD-1, will be combined with pemetrexed+platinum (Investigators choice of cisplatin or carboplatin) chemotherapy to treat participants with advanced or metastatic nonsquamous non-small cell lung cancer (NSCLC) who have not previously received systemic therapy for advanced disease. When the preliminary efficacy and safety data are acquired, a single-blinded phase III study will ensue, in which the efficacy and safety of HX008+pemetrexed+platinum VS pembrolizumab+pemetrexed+platinum in participants of the same population will be compared head-to-head with 1:1 randomization. The primary endpoints are safety and ORR (overall response rate) evaluated by the investigator in phase II study, and PFS evaluated by IRC (independent review committee) in phase III study. The primary hypothesis in phase III study is that HX008+pemetrexed+platinum is non-inferior to pembrolizumab+pemetrexed+platinum in terms of PFS (Progression-Free Survival).

ELIGIBILITY:
Inclusion Criteria:

* Understood and signed an informed consent form.
* Age ≥ 18 years old, male or female.
* Have a histologically or cytologically confirmed diagnosis of stage IV (M1a or M1b- AJCC 7th edition) nonsquamous NSCLC.
* Have not received prior systemic treatment for their advanced/metastatic NSCLC. Subjects who received adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 12 months prior to the development of metastatic disease.
* Have confirmation that EGFR or ALK-directed therapy is not indicated.
* Have at least one measurable lesion according to RECIST1.1. Lesions situated in previously irradiated areas could be considered as target lesions if progression has been demonstrated in such lesions. If measurable lesions exist in other areas, lesions in previous irradiated areas should be considered as non-target lesions.
* Have provided tumor tissue from locations not radiated prior to biopsy for determination of PD-L1 status prior to randomization. Formalin fixed specimens the subject has been diagnosed with metastatic disease will be preferred. Biopsies obtained prior to receipt of adjuvant/neoadjuvant chemotherapy will be permitted if recent biopsy is not feasible.
* Life expectancy ≥ 3 months.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Score.
* Have adequate organ function as indicated by the following laboratory values:

  1. Blood routine: serum albumin ≥2.5g/dL; absolute neutrophil count (ANC) ≥1.5×10^9/L; while blood cell count (WBC) ≥3×10^9/L; platelet count (PLT) ≥100×10^9/L; hemoglobin (HGB) ≥90 g/L (without blood transfusion within 4 weeks prior to enrollment);
  2. Renal function: creatinine clearance (CrCl) ≥50 mL/min;
  3. Liver function: Patients without liver metastases require alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN. Patients with liver metastases require: ALT and AST≤5×ULN. Serum total bilirubin ≤1.5xULN or direct bilirubin ≤ULN for subjects with total bilirubin levels >1.5xULN;
  4. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless the subject is receiving anticoagulant therapy; OR activated Partial Thromboplastin Time (aPTT) or Partial Thromboplastin Time (PTT) ≤1.5 X ULN unless the subject is receiving anticoagulant therapy.
* If female of childbearing potential, have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* If female of childbearing potential, be willing to use an adequate method of contraception as outlined in Section 4.3-Contraception, for the course of the study through 120 days after the last dose of study medication or through 180 days after last dose of chemotherapeutic agents as specified in the protocol. If male subject with a female partner(s) of child-bearing potential, must agree to use an adequate method of contraception as outlined in Section 4.3-Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy or through 180 days after last dose of chemotherapeutic agents as specified in the protocol. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

* Has predominantly squamous cell histology NSCLC. Mixed tumors will be categorized by the predominant cell type; if small cell elements are present, the subject is ineligible.
* Before the first dose of trial treatment:

  1. Has received prior systemic cytotoxic chemotherapy or other antineoplastic therapy (e.g., erlotinib, crizotinib, cetuximab) for metastatic disease
  2. Had major surgery within 3 weeks prior to the first dose of trial treatment
  3. Has participated in other clinical trial within 4 weeks prior to the first dose
  4. Received radiation therapy to the lung that is > 30 Gy within 6 months prior to the first dose
  5. Completed palliative radiotherapy within 7 days prior to the first dose
  6. Has received a live-virus vaccination within 30 days prior to the first dose. Seasonal flu vaccines that do not contain live virus are permitted.
* Has clinically active diverticulitis, intra-abdominal abscess, GI obstruction, peritoneal carcinomatosis.
* Suffered from other malignant tumors in the past 5 years, except those with low risk of metastasis and death (5-year survival rate > 90%), for instance, skin basal cell carcinoma, squamous cell carcinoma, and carcinoma in situ from cervix or other regions that have been adequately treated.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are clinically stable for at least 2 weeks and, have no evidence of new or enlarging brain metastases and also are off steroids 3 days prior to dosing with study medication. Stable brain metastases by this definition should be established prior to the first dose of study medication. Subjects with known untreated, asymptomatic brain metastases (ie, no neurological symptoms, no requirements for corticosteroids, no or minimal surrounding edema, and no lesion >1.5 cm) may participate but will require regular imaging of the brain as a site of disease.
* Has a known sensitivity to macromolecular agents or any component of cisplatin, carboplatin or pemetrexed.
* Has a history of organ or stem-cell transplantation.
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has received systemic corticosteroids (a calculated dose >10mg prednisone per day ) or other immunosuppressive drugs within 14 days before the first administration of the study drug, excluding:

  1. Nasal spray, inhalation or other local glucocorticoids.
  2. Short-term (≤ 7 days) use of glucocorticoids as a preventive medication for allergic reactions or as a therapeutic medication for non-autoimmune diseases.
* Is on chronic systemic steroids. Subjects with asthma that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections would not be excluded from the study.
* Is unable to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs), other than an aspirin dose ≤ 1.3 g per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam).
* Is unable or unwilling to take folic acid or vitamin B12 supplementation.
* Had prior treatment with any anti-PD-1, or PD-L1 or PD-L2 agent or an antibody targeting other immuno-regulatory receptors or mechanisms. Examples of such antibodies include (but are not limited to) antibodies against IDO, PD-L1, IL-2R, GITR.
* Has a severe active infection prior to the first administration of the study drug and might not in the best interest of the subject to participate, in the opinion of the Investigator.
* Has known history of Human Immunodeficiency Virus (HIV) (known HIV 1/2 antibodies positive).
* Has known active Hepatitis B or C. Active Hepatitis B is defined as a known positive HBsAg result. Active Hepatitis C is defined by a known positive Hep C Ab result and known quantitative HCV RNA results greater than the lower limits of detection of the assay. Those with HBV DNA viral load or copy number lower than the lower limits of detection of the assay or HCV RNA negative after adequate treatment is eligible.
* Has known psychiatric or mental disorders, such as epilepsy, dementia, or a known regular user of any illicit drugs, or had a recent history (within the last year) of substance abuse (including alcohol) that would interfere with cooperation with the requirements of the trial.
* Has symptomatic ascites or pleural effusion. A subject who is clinically stable following treatment for these conditions (including therapeutic paracentesis) is eligible.
* Has a history of non-infectious pneumonitis that required steroids or active interstitial pneumonia. Other moderate and severe lung diseases that may interfere with the detection or treatment of study drug-related pulmonary toxicity or seriously affect respiratory function, such as idiopathic pulmonary fibrosis, organic pneumonia / bronchiolitis obliterans, etc (except for local pneumonia induced by radiotherapy).
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
* Has active tuberculosis.
* Has uncontrolled systemic diseases, for instance, cardiovascular and cerebrovascular disease, diabetes, hypertension, etc.
* Has a history or current evidence of any condition, or laboratory abnormality that might not in the best interest of the subject to participate, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-09-25 (Estimated); Study Completion 2023-09-25 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 in phase II study | 12 months
Objective Response Rate (ORR) in phase II study | 12 months
  Percentage of subjects achieving complete response (CR) and partial response (PR)
Progression-Free Survival (PFS) in phase III study | 24 months
  The time from the first study drug treatment to disease progression (PD) or to death of the subject due to any reason.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) in phase III study | 24 months
  The time from the first study drug treatment to disease progression (PD) or to death of the subject due to any reason.
Progression-Free Survival (PFS) in phase II study | 24 months
  The time from the first study drug treatment to disease progression (PD) or to death of the subject due to any reason.
Duration of Response (DOR) in phase II and III study | 24 months
  Duration of Response (DOR) is defined as the time from the first evidence of response (PR or CR) to the first evidence of PD or the date of death for any reason.
12-month PFS rate in phase II and III study | 24 months
  The rate of participants who experienced neither disease progression (PD) nor death due to any reason in one year after the first study drug treatment.
Overall survival (OS) in phase II and III study | 36 months
  Overall survival (OS) refers to the time from the first study drug treatment to death due to any cause.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 in phase III study | 36 months
  Evaluating the safety and tolerance of HX008+pemetrexed+platinum as the first-line treatment in the participants with advanced or metastatic nonsquamous NSCLC.

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Chaoyang Hospital ,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Hunan Province Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Liaoning Cancer Hospital & Insititute, Shenyang, Liaoning
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Affiliated Hangzhou Cancer Hospital, Hangzhou, Zhejiang